CLINICAL TRIAL: NCT05283486
Title: A Double-blind, Randomized, Phase 2 Study to Investigate the Efficacy, Tolerability and Pharmacokinetics of MYMD1 in the Treatment of Participants Aged 65 Years or Older With Chronic Inflammation Associated With Sarcopenia/Frailty
Brief Title: Evaluation of Efficacy, Tolerability, and Pharmacokinetics of MYMD1 for Chronic Inflammation and Sarcopenia/Frailty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TNF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MyMD-PK-003
Record Dates: First submitted 2022-02-16; First posted 2022-03-17 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-03

CONDITIONS: Sarcopenia; Frailty; Aging
Keywords: frailty; aging; sarcopenia
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — isomyosmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: MYMD1 600mg (Experimental): Subjects randomly assigned to the MYMD1 600mg cohort
  Interventions: Drug: MYMD-1 600MG
- Cohort 1: Placebo 600mg (Placebo Comparator): Subjects assigned to the 600mg placebo group
  Interventions: Drug: placebo 600mg
- Cohort 2: MYMD1 750mg (Experimental): Subjects randomly assigned to the MYMD1 750 cohort
  Interventions: Drug: MYMD-1 750mg
- Cohort 2: Placebo 750mg (Placebo Comparator): Subjects assigned to the 750mg placebo group
  Interventions: Drug: placebo 750mg
- Cohort 3: MYMD1 900mg (Experimental): Subjects randomly assigned to the MYMD1 900mg cohort
  Interventions: Drug: MYMD-1 900mg
- Cohort 3: Placebo 900mg (Placebo Comparator): Subjects assigned to the 900mg placebo group
  Interventions: Drug: placebo 900mg
- Cohort 4: MYMD1 1050mg (Active Comparator): Subjects randomly assigned to the MYMD1 1050mg cohort
  Interventions: Drug: MYMD-1 1050mg
- Cohort 4: Placebo group 1050mg (Placebo Comparator): Subjects assigned to the 1050mg placebo group
  Interventions: Drug: placebo 1050mg

INTERVENTIONS:
Drug: MYMD-1 600MG — Cohort 1: 600mg drug
  Other Names: MYMD1 600mg
  Arms: Cohort 1: MYMD1 600mg
Drug: MYMD-1 750mg — Cohort 2: 750mg drug
  Other Names: MYMD1 750mg
  Arms: Cohort 2: MYMD1 750mg
Drug: MYMD-1 900mg — Cohort 3: 900mg drug
  Other Names: MYMD1 900mg
  Arms: Cohort 3: MYMD1 900mg
Drug: MYMD-1 1050mg — Cohort 4: 1050mg drug
  Other Names: MYMD1 1050mg
  Arms: Cohort 4: MYMD1 1050mg
Drug: placebo 600mg — Cohort 1: 600mg placebo
  Other Names: placebo-600mg
  Arms: Cohort 1: Placebo 600mg
Drug: placebo 750mg — Cohort 2: 750mg placebo
  Other Names: placebo-750mg
  Arms: Cohort 2: Placebo 750mg
Drug: placebo 900mg — Cohort 3: 900mg placebo
  Other Names: placebo-900mg
  Arms: Cohort 3: Placebo 900mg
Drug: placebo 1050mg — Cohort 4: 1050mg placebo
  Other Names: placebo-1050mg
  Arms: Cohort 4: Placebo group 1050mg

SUMMARY:
The study will be conducted to investigate the efficacy, tolerability and pharmacokinetics of MYMD1 in participants with chronic inflammation associated with sarcopenia/frailty, a condition linked to elevated levels of proinflammatory cytokines.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled evaluation of the efficacy, tolerability and pharmacokinetics (PK), of MYMD1 in participants aged 65 years or older with chronic inflammation associated with sarcopenia/frailty. After participants sign the informed consent form (ICF), they will enter the screening period which will not exceed 28 days. Participants who fulfill all the inclusion criteria and none of the exclusion criteria will be randomized (4:1) to receive MYMD1 or placebo in a blinded fashion until the end of-study (EOS) visit on Day 28. A participant is considered to have completed the study if he/she has completed all phases of the study including the EOS visit scheduled on Day 28.

Follow up: Participants will be contacted within 24 hours post Day 1 treatment for routine medical assessment. Participants will be contacted by phone every two days post discharge until day 7 visit. Week two post discharge participants will be instructed to call the Clinical nurse and/or the 24-hour medical monitor for any study related concerns. After the EOS visit, participants will be contacted by phone weekly for a completed 30 day follow up and documented close out.

Study treatment will be dispensed on Day 1 of each cohort. Cohort 1 will be required to take 600mg [4 capsules of 150 mg each or matching placebo]; Cohort 2 will be required to take 750mg ([5 capsules of 150 mg each or matching placebo]; Cohort 3 will be required to take 900mg ([6 capsules of 150 mg each or matching placebo]; and Cohort 4 will be required to take 1050mg ([7 capsules of 150 mg each or matching placebo] orally each orally each day throughout the treatment duration.

On Day 1, a single, oral dose of MYMD1 or placebo will be administered following an overnight fast of at least 12 hours. The participants may have applesauce, 15 to 20 minutes post dose.

Number of Investigators and Study Centers:

Approximately 2 sites are expected to participate in this study.

Number of Participants:

Approximately 40 participants will be enrolled in this study; 32 participants will receive the study treatment (MYMD1) and 8 will receive the placebo.

Treatment Groups and Duration:

The overall duration for all participants enrolled in this study will be 28 days. Serial PK sampling will be collected across all cohorts.

Statistical methods:

Incidence of adverse events will be summarized by dose level, by preferred term, and by severity and relationship to the study treatment.

Descriptive statistics will be tabulated for clinical laboratory tests, electrocardiogram intervals, and vital signs.

MYMD1 concentrations and calculated PK parameters will be summarized by dose level and study data. Dose proportionality of MYMD1 will be explored graphically, and if appropriate, by using a regression model.

Pyridyloxobutyl and tumor necrosis factor-α results and corresponding changes from baseline will be summarized by dose level.

Individual participant data will be presented in listings.

For change from baseline efficacy analyses, only participants with a baseline and at least one non missing postbaseline measurement will be included.

Treatment emergent Adverse Eventss (TEAEs) by maximum severity, TEAEs by relationship to study treatment, Serious Adverse Events, TEAEs leading to death, and TEAEs leading to discontinuation of study treatment will be tabulated for each treatment group. Commonly occurring TEAEs in either treatment group, will be summarized using descriptive statistics.

All laboratory test results, vital signs measurements, electrocardiogram (ECG) results, and weight will be summarized for each treatment group using descriptive statistics at each visit for raw numbers and change from baseline. The incidence of treatment emergent abnormal laboratory values, vital signs, neurological exam and ECG values will also be summarized using descriptive statistics.

Safety Review Committee A Safety Review Committee (SRC) consisting of the Investigator, Medical Monitor, and PK Scientist will review the available PK safety data to decide whether to escalate to the next higher planned dose, to repeat a dose level or to stop the dose escalation. To maintain the treatment assignment blinded, safety data will exclude treatment assignment and PK data will have blinded participant identification numbers. All SRC decisions, along with their rationale, will be documented in writing, and retained in the study files.

The data review and analysis will be based on the available Investigator-reported data in the clinical database at that time. Data to be reviewed will include safety, tolerability, and available PK data through day 8.

The Coordinating Investigator and the Sponsor, when appropriate, will invite other specialist individuals to participate in the review, eg, PK scientists, statisticians, and clinical specialists. MyMD Pharmaceuticals, Inc. will also have a board-certified cardiologist and neurologist available for consultation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 years or older, at the time of signing the ICF

   Type of Participant and Disease Characteristics
2. Elevated biomarkers of inflammation (serum IL-6 level ≥2.5 pg/mL and/or sTNFR1 level ≥1500 pg/mL)
3. Low gait speed ≤ 0.8 m/s
4. Short Physical Performance Battery (SPPB) score ≤8

   Weight
5. Body weight ≥35 kg Other
6. Adequate dietary intake
7. Able to complete a 4-meter timed walk
8. Assessment and documentation of sarcopenia-related loss of muscle mass based on Dual-energy X-ray absorptiometry (DXA) -derived appendicular skeletal muscle mass index (ASMI) measurements.

   Reproductive Status
9. Male participants who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
10. Female participants are eligible to participate if they do not qualify as a woman of childbearing potential (WOCBP)

    Informed Consent
11. Capable of giving signed informed consent as described in Appendix 2, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol

Exclusion Criteria:

1. Taking anti-inflammatory drugs on a daily basis. Note: If the participant has been stable on their antidepressant regimen for at least 3 months and agrees not to increase the medicine for the 28 days of treatment in the trial, they may be allowed into the study
2. Currently tobacco users or those who used tobacco within 30 days of study entry
3. Dementia, encephalopathy or any medical condition impacting cognition
4. Medical conditions that would impact mobility testing or handgrip strength including
5. Rheumatoid arthritis, any autoimmune condition, Parkinson's disease, muscular dystrophy, cerebral vascular accident, lower or upper extremity neuropathy, major skeletal joint deformity, upper extremity joint dysfunction, partial or complete upper extremity amputation or missing anatomy impacting grip, history of pain with walking, gout, chronic obstructive pulmonary disease, congestive heart failure, exercise induced angina, lower extremity amputation (partial or complete) or missing anatomy impacting walking, recent surgery or hospitalization (past 3 months); lower or upper extremity fracture in the past 6 months, lower or upper extremity tendinitis, diagnosis of cancer other than basal cell carcinoma, dialysis dependent renal disease, Meniere's disease, spinal cord fracture or compression, paraplegia or quadriplegia or any other medical condition that in the opinion of the Investigator would impair measurement of a 6-minute walk or handgrip strength
6. A lower limb fracture in the past 6 months or any impairment or disease severely affecting gait (eg, stroke with hemiparesis, myasthenia gravis, Parkinson's disease, peripheral polyneuropathy, intermittent claudication in advanced peripheral vascular disease, spinal stenosis, or severe osteoarthritis of the knee or hip with ineffective pain management)
7. Requires regular assistance from another person for general activities of daily living (eg, bathing, dressing, toileting)
8. History of cardiac conduction abnormalities, arrhythmias, and/or bradycardia
9. Intraocular surgery and laser procedures for refractive correction within 6 months prior to screening
10. Any underlying muscle disease including active myopathy or muscular dystrophy
11. Confirmed diagnosis of heart failure classified as New York Heart Association Class III or IV (eg, dilated cardiomyopathy)
12. Type I diabetes or uncontrolled Type 2 diabetes
13. Chronic kidney disease (estimated glomerular filtration rate [eGFR] <60 mL/min)
14. History of confirmed chronic obstructive pulmonary disease with a severity Grade >2 on the Medical Research Council Dyspnea Scale
15. Confirmed rheumatoid arthritis or other systemic autoimmune disease requiring immunosuppressive therapy or corticosteroids >10 mg/day prednisone equivalent
16. Known history or presence of severe active acute or chronic liver disease (eg, cirrhosis)
17. Myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention (eg, angioplasty or stent placement), or deep vein thrombosis/pulmonary embolism within 12 weeks of screening
18. Active cancer (ie, under current treatment), or cancer requiring treatment in the last 5 years excluding non-melanoma skin cancers or cancers with excellent prognosis (eg, early-stage prostate or breast cancer, carcinoma in situ of the uterine cervix)
19. Any known chronic active infection
20. Use of any anxiolytics, cannabis or opioid medications
21. Currently abusing drugs or alcohol, and/or have a history of drug or alcohol dependence within 6 months of entering this study
22. A score of <23 on the Mini Mental Status Exam
23. Treatment with any prescription or investigational drugs, devices or chemotherapy, or any other therapies for sarcopenia
24. Use of medications with narrow therapeutic ranges within 48 hours of the first dose of study treatment
25. Current use of systemic steroids or use of systemic steroids within 90 days of treatment except for prophylaxis against imaging contrast dye allergy or replacement-dose steroids in the setting of adrenal insufficiency (providing this is ≤10 mg/day prednisone or equivalent; see Appendix 5 for steroid conversion table), or transient exacerbations of other underlying diseases such as chronic obstructive pulmonary disease requiring treatment for <3 weeks
26. Vaccination with live vaccines while on study

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Demonstrate reduction of chronic inflammatory markers in participants treated with MYMD1 | Screening
  Effect on serum levels of sTNFR1, IL-6, and TNFα over 28 days of treatment
Demonstrate reduction of chronic inflammatory markers in participants treated with MYMD1 | Day 1
  Effect on serum levels of sTNFR1, IL-6, and TNFα over 28 days of treatment
Demonstrate reduction of chronic inflammatory markers in participants treated with MYMD1 | Day 7
  Effect on serum levels of sTNFR1, IL-6, and TNFα over 28 days of treatment
Demonstrate reduction of chronic inflammatory markers in participants treated with MYMD1 | Day 14
  Effect on serum levels of sTNFR1, IL-6, and TNFα over 28 days of treatment
Demonstrate reduction of chronic inflammatory markers in participants treated with MYMD1 | Day 21
  Effect on serum levels of sTNFR1, IL-6, and TNFα over 28 days of treatment
Demonstrate reduction of chronic inflammatory markers in participants treated with MYMD1 | Day 28
  Effect on serum levels of sTNFR1, IL-6, and TNFα over 28 days of treatment
To evaluate the PK of oral doses of MYMD1 capsules | Cohorts 1, 2, 3, 4: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24 hrs; Day 7, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24; Day 14, pre-dose, 0.5 hrs; Day 21, pre-dose, 0.5 hrs; Day 28, pre-dose, 0.5 hrs]
  Area Under the Curve (AUC) (0-last): variation of a drug concentration in blood plasma as a function of time, compared across treatment and placebo groups.
To evaluate the PK of oral doses of MYMD1 capsules | Cohorts 1, 2, 3, 4: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24 hrs; Day 7, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24; Day 14, pre-dose, 0.5 hrs; Day 21, pre-dose, 0.5 hrs; Day 28, pre-dose, 0.5 hrs]
  Pharmacokinetics: Cmax - Maximum Concentration of drug substance in blood plasma, compared across treatment and placebo groups.
To evaluate the PK of oral doses of MYMD1 capsules | Cohorts 1, 2, 3, 4: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24 hrs; Day 7, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24; Day 14, pre-dose, 0.5 hrs; Day 21, pre-dose, 0.5 hrs; Day 28, pre-dose, 0.5 hrs]
  Pharmacokintetics: tmax - Time to Maximum Concentration of drug substance in blood plasma, compared across treatment and placebo groups.
To evaluate the PK of oral doses of MYMD1 capsules | Cohorts 1, 2, 3, 4: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24 hrs; Day 7, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24; Day 14, pre-dose, 0.5 hrs; Day 21, pre-dose, 0.5 hrs; Day 28, pre-dose, 0.5 hrs]
  Pharmacokinetics: t1/2 - Time to metabolize 1/2 of dose (eg, half-life) of drug substance, measured in blood plasma, compared across treatment and placebo groups.
To evaluate the PK of oral doses of MYMD1 capsules | Cohorts 1, 2, 3, 4: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24 hrs; Day 7, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24; Day 14, pre-dose, 0.5 hrs; Day 21, pre-dose, 0.5 hrs; Day 28, pre-dose, 0.5 hrs]
  Pharmacokinetics: CL/F - Oral Clearance of the drug substance (CL/F), compared across treatment and placebo groups.
To evaluate the PK of oral doses of MYMD1 capsules | Cohorts 1, 2, 3, 4: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24 hrs; Day 7, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 24; Day 14, pre-dose, 0.5 hrs; Day 21, pre-dose, 0.5 hrs; Day 28, pre-dose, 0.5 hrs]
  Pharmacokinetics: Volume of Distribution (V2/F ) - Volume of Distribution of the drug substance (V2/F), compared across treatment and placebo groups.
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 1 (predose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 1 (0-4 hrs post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 1 (4-8 hrs post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 1(8-24hrs post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 7 (predose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 7 (0-4 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 7 (4-8 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 7 (8-24hrs post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 14 (predose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 14 (0-4 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 14 (4-8 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 14 (8-24 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 21 (predose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK of oral doses of MYMD1 capsules | Day 21 (0-4 hrs post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 21 (4-8 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 21 (8-24 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 28 (pre dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 28 (0-4hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 28 (4-8 hours post dose)
  urine sample collection for presence of parent drug - MYMD1
To evaluate the PK (urine) of oral doses of MYMD1 capsules | Day 28 (8-24 hours post dose)
  urine sample collection for presence of parent drug - MYMD1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Dunn, MD, Principal Investigator — Clinical Research of West Florida; Lon Lynn, DO, Principal Investigator — Clinical Research of West Florida; Jeremy Walston, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No